CLINICAL TRIAL: NCT02881359
Title: SEAL Registry - Observational, Retrospective and Prospective, One Arm, Registry Study for the Effectiveness of LifeSeal® Kit on Anastomotic Leaks in Patients Undergoing Low and Ultralow Anterior Resection
Brief Title: SEAL Registry - European Registry for the Effectiveness of LifeSeal® Kit
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: LifeBond Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-LS-0146
Record Dates: First submitted 2016-08-23; First posted 2016-08-29 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Anastomotic Leakage
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LifeSeal® Kit: creation of a coloanal or colorectal anastomosis
  Interventions: Device: LifeSeal® Kit

INTERVENTIONS:
Device: LifeSeal® Kit — used as an adjunct to suture or staple line during standard surgical repair of the GI tract (anastomosis or linear) to provide re-inforcement and help reduce leaks.

SUMMARY:
This study will assess the effectiveness of commercially available LifeSeal® Kit as measured by the incidence of post-operative clinical anastomotic leak rates in subjects undergoing low and ultralow anterior resection with an anastomosis. All patients treated with LifeSeal® will be offered to participate

DETAILED DESCRIPTION:
The LifeSeal® Kit is a novel surgical sealant intended to be used as an adjunct to suture or staple line during standard surgical repair of the GI tract (anastomosis or linear) to provide re-inforcement and help reduce leaks. The LifeSeal™ Kit has recently been CE certified on March 2016 for marketing in the European Union.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at screening visit
2. Written informed consent obtained
3. Subject is scheduled to have or already underwent elective open, laparoscopic or robot assisted surgery involving the creation of a coloanal or colorectal anastomosis* created within 15 cm from the anal verge.
4. Subject was already treated or is scheduled to be treated with LifeSeal® Kit, applied according to the IFU

Exclusion Criteria:

1. Subject with American Society of Anesthesiology (ASA) status > 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are treated with LifeSeal® and comply with the eligibility criteria will be offered to participate in the study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-08 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-operative clinical anastomotic leaks at discharge | discharge from hospital 3-14 days post surgery

SECONDARY OUTCOMES:
Incidence of post-operative clinical anastomotic leaks up to 4 weeks post-surgery | up to 4 weeks post surgery

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (7):
  - Algemeen Stedelijk Ziekenhuis, Aalst
  - ZNA Antwerpen Campus, Antwerp
  - Jessa Ziekenhuis, Hasselt
  - Jan Yperman Ziekenhuis, Ieper
  - CHR de la Citadelle, Liège
  - H. Hartziekenhuis, Mol
  - AZ Delta, Roeselare
- ZGT, Almelo, Netherlands

IPD SHARING:
Plan to Share IPD: No